CLINICAL TRIAL: NCT03526614
Title: REpetitive Assessement of Thromboembolic and Bleeding SCOREs in Patients Treated With Dual Antiplatelet Therapy
Brief Title: REpetitive Assessement of SCOREs in Patients on Dual Antiplatelet Therapy
Acronym: RE-SCORE
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Other Study IDs: 2018/D/401
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Dual Anti-platelet Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients treated with percutaneous coronary intervention (PCI) require dual antiplatelet therapy (DAPT). Preliminary assessment of the PRECISE-DAPT score is mandatory in order to assess the risk of bleeding while on DAPT. The score takes into consideration age, creatinine clearance, haemoglobin, white-blood-cell count and previous spontaneous bleeding. One should consider, however, that some of the variables included in the PRECISE-DAPT score might change with time. As a consequence, the PRECISE-DAPT score should not be considered a static score as it might vary after the initial computation. It remains unknown, however, if the delta PRECISE-SCORE, reflecting the change in score between baseline and follow-up, might predict more reliably the long-term bleeding risk of PCI patients.

DETAILED DESCRIPTION:
The RE-SCORE registry is a multicenter study aimed at comparing the predictive value of the PRECISE-DAPT score assessed at time of discharge vs. the Delta PRECISE-DAPT score, as assessed every 3 months in PCI patients receiving DAPT.

The primary end-point of the study is the occurrence of bleeding, as defined according to the criteria of the Bleeding Academic Research Consortium (BARC), either in the whole study population or in men vs women.

ELIGIBILITY:
Inclusion Criteria: All patients undergoing percutaneous coronary intervention and treated with dual antiplatelet therapy for at least 3 months

Exclusion Criteria: Contraindications to dual antiplatelet therapy lasting more than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease and indication to PCI
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Bleeding in the overall population | Up to 12 months
  Bleeding episodes
Bleeding in men and women | Up to 12 months
  Bleeding episodes

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, Study Chair — University of Roma La Sapienza
Locations (1):
- University Sapienza, Rome, Please Select, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pelliccia F, Gragnano F, Pasceri V, Marazzi G, Cacciotti L, Placanica A, Niccoli G, Palmerini T, Speciale G, Granatelli A, Calabro P. Gender-related differences in changes of estimated bleeding risk in patients on dual antiplatelet therapy: the RE-SCORE multicenter prospective registry. Platelets. 2022 Nov 17;33(8):1228-1236. doi: 10.1080/09537104.2022.2102602. Epub 2022 Jul 25. PMID 35875853
- [Derived] Pelliccia F, Pasceri V, Marazzi G, Cacciotti L, Placanica A, Gragnano F, Niccoli G, Palmerini T, Tanzilli G, Speciale G, Granatelli A, Calabro P, Crea F, Gaudio C. Predictive ability of longitudinal changes in PRECISE-DAPT score in patients on dual antiplatelet therapy: The RE-SCORE multicentre prospective registry. Eur J Prev Cardiol. 2021 Oct 13;28(12):e36-e38. doi: 10.1177/2047487320937846. Epub 2020 Jul 5. No abstract available. PMID 34647586